CLINICAL TRIAL: NCT00910325
Title: Natural Orifice Translumenal Endoscopic Surgery: Laparoscopic-Assisted Transvaginal Cholecystectomy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The alternative laparoscopic chole, has so little morbidity very few patients opt for a transvaginal approach when presented with the alternative
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David W. Rattner, MD, Chief, Division of General and Gastrointestinal Surgery, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008p001938
Record Dates: First submitted 2009-05-27; First posted 2009-05-29 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Cholelithiasis
Keywords: Female; Cholelithiasis; Natural Orifice Surgery; Laparoscopic- Assisted; Transvaginal
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Laparoscopic-assisted transvaginal cholecystectomy — Trans-vaginal Cholecystectomy with Laparoscopic Assistance

SUMMARY:
To determine the feasibility, safety, and efficacy of a novel minimally invasive approach to cholecystectomy and to establish a description of this novel translumenal technique in humans at this institution.

ELIGIBILITY:
Inclusion Criteria:

* Females who are postmenopausal or who no longer wish to bear children
* Females >25 years old and <65 years old
* Diagnosis of biliary disease requiring cholecystectomy
* American Society of Anesthesiology (ASA) Class I or II
* Females who are able to understand and willing to sign an informed consent document

Exclusion Criteria:

* Pregnancy
* BMI >= 30
* Patients who are still interested in childbearing
* Patients taking immunosuppressive medications or who are immunocompromised
* Patients with acute cholecystitis or history of acute cholecystitis ( as defined by right upper quadrant pain with history of fevers and/or elevated white blood cell count and/or positive ultrasound findings, ie, gallbladder wall thickening or pericholecystic fluid)
* Patients with suspicion of gallbladder cancer
* Patients with history of previous open abdominal surgery
* Patients with untreated common bile duct stones

Ages: 26 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2008-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The safety and efficacy of the procedure | one year

SECONDARY OUTCOMES:
Post-operative pain | one year
Time to return to work | one year
Time to return to daily activities | one year

CONTACTS AND LOCATIONS:
Overall Officials: David W Rattner, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States